CLINICAL TRIAL: NCT05391685
Title: EFFECT OF SCAR RELEASE TECHNIQUES ON CHRONIC SCAR PAIN AND MOBILITY POST CESAREAN SECTION
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nabiha Mahmoud Ahmed Mahmoud, Specialist of physical therapy at Elmansoura International hospital, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/003710
Record Dates: First submitted 2022-05-21; First posted 2022-05-26 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Cesarean Section Complications
MeSH Terms: interventions — Ultrasonic Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- therapeutic ultrasound (Experimental): Control group will be treated by therapeutic ultrasound only
  Interventions: Other: Scar release techniques + therapeutic ultrasound
- therapeutic ultrasound+scar release techniques (Experimental): Study group will be treated by various scar release techniques in addition to therapeutic ultrasound
  Interventions: Other: Scar release techniques + therapeutic ultrasound

INTERVENTIONS:
Other: Scar release techniques + therapeutic ultrasound — Control group will be treated by therapeutic ultrasound only for2 sessions per week for two weeks Study group) will be treated by various scar release techniques in addition to therapeutic ultrasound, 2 sessions per week for two weeks.

SUMMARY:
Purpose of the study:

The aim of this study is to determine the effect of scar release techniques on chronic scar pain and mobility post cesarean section.

Hypothesis:

* H0: There is no effect of scar release techniques on chronic scar pain and mobility post cesarean section.
* HA: There is effect of scar release techniques on chronic scar pain and mobility post cesarean section.

DETAILED DESCRIPTION:
A vicious impediment on quality of life including psychological and functional disability, and interference with baby care and bonding may occur among women who experience chronic post-caesarean section pain (CPCSP) .

Structural alterations of the skin and subcutaneous tissues with scarring result in reduced mobility and viscoelasticity that could cause compression of the sensory receptors and nerve ﬁbers and disrupt their signaling. The viscoelastic properties could potentially be modiﬁed when the skin and scars are stressed and/or strained by manual therapies and this can affect the sensitivity threshold of the mechanosensitive and nociceptive receptors.

There are limited studies about the effect of various scar release techniques on chronic post cesarean section scar pain and mobility and their impact on quality of life on the affected women . So, this study will be helpful and of valuable benefits for medical services organizations and increase body of knowledge of physical therapists in scientific field.

This study will be conducted on forty women suffering from chronic post cesarean section scar pain and restricted scar mobility , they will be referred from department of Obestetrics and Gynaecology in Elmansoura International Hospital, Egypt.

ELIGIBILITY:
Inclusion Criteria:

* Women with a well healed, old , transverse cesarean section scar (more than 6 months resulted in chronic scar pain).
* Pain can be intermittent or constant at rest or with activity, and it is reported to be at least at a level of about 3/ 10 on visual analogue scale at recording sites will be marked on the C-section scar at 2.5 cm intervals .
* Women identified that the pain is either located in the cesarean section scar or caused by palpation of scar and it presents since the time of surgery not prior to the cesarean section.
* Their ages will range from 25-35 years old.
* Their BMI will be 18.5-29.9 kg/ m².
* Voluntary acceptance to participate in the study.

Exclusion Criteria:

* Women will be excluded if they have :
* Acute and subacute cesarean section.
* Delayed wound healing.
* History of abdominal or pelvic cancer.
* Active pelvic or abdominal infection.
* Skin irritation/inflammation at the site of scar.
* Currently pregnant women.

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-06-20 (Estimated); Primary Completion 2022-09-20 (Estimated); Study Completion 2022-10-20 (Estimated)

PRIMARY OUTCOMES:
pain intensity | up to 4 weeks
  The pain intensity will be assessed through visual analouge scale( VAS )for all participating women in both groups before and after the end of the treatment program. Each woman will be asked to mark a point on the line between the extremes that is related to her pain intensity.
Pressure pain threshold | up to 4 weeks
  A pressure algometer will be used to measure pressure pain threshold (PPT)for all participating women in both groups before and after the end of the treatment program.
  PPT recording sites will be marked on the C-section scar at 2.5 cm intervals. This resulted in from 5 to 8 measurement points along the scar.
  Following, the marked points will be used to record PPTs in all time points for the PPT assessment; a 1-cm2 pressure probe will be positioned perpendicularly to the skin and pressed at a rate of 30kPa/s.Two measures will be collected for each area, with 30 second rest between point testing.
  Average pressure pain threshold (AvPPPT) (pressure points across worst 3 points on scar averaged) will be used for the analysis of the PPT data
Patient and Observer Scar Assessment Scale (POSAS) | up to 4 weeks
  It will be used pre and post- treatment to assess the symptoms of pain and pruritus at the cesarean section scar for all participanting women of both groups before and after the end of the treatment program.
Scar adherence | up to 4 weeks
  post cesarean section scar adherence will be assessted by an adheremeter for both groups before and after the end of treatment program.
  A mark will be made on the tightest part of the scar in four directions (superior, inferior, right and left). As there is no a contralateral side to abdominal tissue to be used as a reference range, we will use multi-directional scar mobility (MDM) .
  Scar mobility measurements across the points will be averaged for each participating women .

SECONDARY OUTCOMES:
Quality of life | up to 4 weeks.
  SF-36 questionnaire will be used to assess the health related quality of life for all women in both groups before and after the end of the treatment program.

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF